CLINICAL TRIAL: NCT06322641
Title: FLAME-ASCVD-Nephro A Multinational Survey-based Study to Understand the Real-world Awareness and Perceptions of Systemic inFLAMmation and rolE of hsCRP as a Biomarker in Patients With AtheroSclerotic CardioVascular Disease and Chronic Kidney Disease Among Nephrologists
Brief Title: A Study to Understand the Real-world Awareness and Perceptions of Systemic inFLAMmation and rolE of hsCRP as a Biomarker in Patients With AtheroSclerotic CardioVascular Disease and Chronic Kidney Disease Among Nephrologists
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8092; U1111-1303-3089 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Chronic Kidney Disease (CKD); Systemic Inflammation
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nephrologist: Nephrologist with ASCVD and CKD patients
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this survey is to collect information for scientific research and to better understand the role of systemic inflammation in identification, treatment and management of patients with Atherosclerotic Cardiovascular Disease (ASCVD) and Chronic Kidney Disease (CKD)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Is a Nephrologist.
* Has been in practice greater than or equal to 3 years.
* Sees at least 20 patients with ASCVD and CKD per month.
* Treats patients for more than only dialysis

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Does not meet inclusion criteria requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nephrologist with ASCVD and CKD patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Nephrologists' perceptions towards the role of systemic inflammation in the identification, treatment and management of patients with ASCVD and CKD | At the time of survey response (Day 1)
  Multi-select from a defined list; Numerical; A 7-point Likert scale for measurement of agreement from 1 "strongly disagree" to 7 "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- KJT Group, Inc., Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com